CLINICAL TRIAL: NCT05701982
Title: The Effect of a Technology-Mediated Integrated Walking and Tai Chi Intervention on Physical Function in Veterans With COPD and Chronic Musculoskeletal Pain
Acronym: WATCH for Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F4225-R
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: COPD; Chronic Musculoskeletal Pain
Keywords: physical activity; mindful movement; videoconference
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention is ESC-TC which is delivered remotely. It a web-based platform (Every Step Counts) to promote walking combined with pain management content, an online Tai Chi video library, and synchronous Tai Chi classes led by an instructor via teleconference. The investigators will randomize participants 1:1 to ESC-TC or usual care for 6 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and study staff who conduct follow-up visits for outcome assessments will be blinded to each participant's randomization group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Every Step Counts-Tai Chi (Experimental): The intervention is ESC-TC which is a web-based platform (Every Step Counts) to promote walking combined with pain management content, an online Tai Chi video library, and synchronous Tai Chi classes led by an instructor via teleconference. The intervention is delivered remotely.
  Interventions: Behavioral: Every Step Counts-Tai Chi
- Usual Care (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Every Step Counts-Tai Chi — The intervention is ESC-TC which is a web-based platform (Every Step Counts) to promote walking combined with pain management content, an online Tai Chi video library, and synchronous Tai Chi classes led by an instructor via teleconference. The intervention is delivered remotely.
  Arms: Every Step Counts-Tai Chi
Other: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
Persons with COPD benefit from being physically active, but they are often limited by chronic musculoskeletal pain. This project will determine whether a non-pharmacologic, integrated, technology-mediated walking and Tai Chi mindfulness intervention can improve physical function in Veterans with COPD and chronic musculoskeletal pain. The proposed research addresses VA Rehabilitation R&D Service's high priority area of improving health-related quality of life by reducing disease burden and maximizing function in Veterans with chronic disease.

DETAILED DESCRIPTION:
Current physical activity (PA) interventions for persons with chronic obstructive pulmonary disease (COPD) focus primarily on reducing the debilitating symptom of dyspnea, or shortness of breath. However, over half of patients with COPD experience chronic musculoskeletal pain which limits achievement of PA goals and optimization of physical function. Low PA is associated with poor outcomes-increased risk of COPD acute exacerbations, hospitalizations, and death-independent of lung function. Funded by Rehabilitation R&D, the investigators have developed Every Step Counts (ESC), a web-based intervention to promote PA in Veterans with COPD. ESC couples a dynamic website with a pedometer that objectively monitors daily step counts. Based on the Behavioral Theory of Self-Regulation, the website provides individualized step-count goals, iterative feedback, education on disease self-management, motivation, and an online community of social support. In RCTs, the investigators have demonstrated ESC's safety, feasibility, and efficacy to increase PA over 3-6 months. However, not all participants increased daily step counts. In secondary analyses, the investigators identified pain as a significant barrier to PA. Participants with co-occurring pain and dyspnea walked 1,200-1,400 fewer steps per day, compared to those with no symptoms. In its current form, ESC does not focus on pain management. Tai Chi (TC) is an attractive nonpharmacologic treatment for chronic musculoskeletal pain. TC improves neuromuscular function, core strength, and lower limb proprioception. Importantly, the mindfulness embedded in TC uniquely addresses cognitive and psycho-emotional processes critical for pain management (i.e., "extinction of fear conditioning, acceptance-based coping strategies, increased ability to self-regulate affective appraisal of nociceptive input," and reduced pain-related distress and catastrophizing). The investigators have shown that persons with COPD can safely engage with TC delivered via either in-person classes or video instruction. The investigators propose to integrate ESC and TC to target biopsychosocial mechanisms of pain to break the chronic pain cycle and improve physical function in persons with COPD. The investigators will adapt ESC with pain management content, an online TC video library, and synchronous TC classes led by an instructor via teleconference. The investigators will randomize participants 1:1 to ESC-TC or usual care for 6 months. Assessments of outcomes will occur at baseline, 2, 4, and 6 months in all participants, and at 12 months in a subset who enroll early. Aim 1: Determine the efficacy of the ESC-TC intervention in 136 persons with COPD and chronic musculoskeletal pain to improve the primary outcome of physical function, measured by daily step count, compared to usual care at 6 months. Aim 2: Evaluate the effect of the ESC-TC intervention on secondary outcomes of (a) pain intensity and interference, (b) dyspnea, (c) health-related quality of life, (d) mobility, (e) depression, (f) exercise self-efficacy, (g) kinesiophobia, (h) pain catastrophizing, and (i) sleep quality. Aim 3: Explore the long-term effects of ESC-TC on symptoms and risk of acute exacerbations and COPD-related hospitalizations at 12 months in approximately 96 participants. The innovative multimodal, web-based, non-pharmacologic intervention to treat chronic musculoskeletal pain has potential to expand access to exercise as a rehabilitation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, aged 40 and older
* Clinical diagnosis of COPD defined as history of cigarette consumption of > 10 pack-years, and either a ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) < 0.70 or chest computerized tomography (CT) evidence of emphysema*
* Numeric Rating Scale pain score > 3 for > 3 months
* Self-reported ability to walk a minimum of one block, bend at the hip, and transfer weight from one leg to another
* Ability to complete 800 feet walk with Fitbit Inspire-2 recording > 90% accuracy to detect steps compared to manual counts*
* Have access to a computer or smartphone with Internet connection or willing to come to study site to use study computers
* Have access to videoconferencing audio and video capabilities
* Competent to provide informed consent and willingness to make return study visits

  * Different criteria are used if baseline study visit is a virtual one.

Exclusion Criteria:

* COPD exacerbation in the previous 1 month
* Clinical signs of unstable cardiovascular disease (active coronary artery disease, congestive heart failure, uncontrolled atrial fibrillation, or uncontrolled hypertension)
* Oxygen saturation < 85% recorded on baseline 4-meter walk*
* High fall risk (unable to perform 5 chair stand tests)
* Inability to ambulate
* Inability to complete questionnaires
* Inability to collect at least 7 of 10 days of baseline step counts
* Active substance abuse
* Participation in a regular exercise (i.e., MOVE! or Gerofit) or Tai Chi program in the previous 3 months
* Concurrent participation in another interventional research study
* Receipt of hospice or end-of-life palliative care
* Active medical intervention that would cause a meaningful increase in pain such as surgery, chemotherapy, or radiation therapy

  * Different criteria are used if baseline study visit is a virtual one.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function measured by Daily Step Counts | 6 months
  The FitBit pedometer will objectively-measure physical activity as daily step counts.

SECONDARY OUTCOMES:
Pain Intensity | 6 months
  The 11-point Numeric Rating Scale (0=no pain; 10=worst pain imaginable) will assess pain intensity.
Dyspnea | 6 months
  Dyspnea will be assessed using the mMRC scale (responses 0-4 with 4 being the most dyspneic).
Pain Interference | 6 months
  The Interference subscale of the West Haven-Yale Multidimensional Pain Inventory will assess pain-related interference, with higher scores representing greater interference.
Dyspnea | 6 months
  UCSD Shortness of Breath Questionnaire with 24 items. Scores range from 0 to 120.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L. Moy, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A Final De-identified, Anonymized Dataset will be created and shared upon request.